CLINICAL TRIAL: NCT04005534
Title: US-Guided Preemptive Brachial Plexus Blockade May Reduce Post-operative Pain: a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CAAE 09012419.3.0000.5501
Record Dates: First submitted 2019-06-24; First posted 2019-07-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain; Rotator Cuff Injuries
Keywords: Postoperative pain; Rotator cuff injuries; Preemptive analgesia
MeSH Terms: conditions — Pain, Postoperative; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective, double-blind and randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each step of the study will be performed by anesthesiologist who will not participate in any other step. All of them, and the patient will be blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Placebo Comparator): Patients from this group will undergo only ultrasound examination of the brachial plexus, two days before the surgery. On the day of surgery they will undergo ultrasound-guided brachial plexus blockade (interscale access; 15 ml 1% ropivacaine and sedation (midazolam 3 mg, fentanyl 50 µg and 15 mg ketamine.
  Interventions: Drug: Standard group
- Preemptive group (Experimental): Patients from this group will undergo ultrasound-guided brachial plexus blockade, two days before the surgery. On the day of surgery they will undergo ultrasound-guided brachial plexus blockade (interscale access; 15 ml 1% ropivacaine and sedation (midazolam 3 mg, fentanyl 50 µg and 15 mg ketamine.
  Interventions: Drug: Preemptive group

INTERVENTIONS:
Drug: Standard group — Ultrasound examination of the brachial plexus 2 days before the surgery. Ultrasound guided brachial plexus blockade and sedation on the day of surgery.
  Other Names: Ultrasound examination
  Arms: Standard group
Drug: Preemptive group — Ultrasound guided brachial plexus blockade 2 days before the surgery. Ultrasound guided brachial plexus blockade and sedation on the day of surgery.
  Other Names: Ultrasound guided blockade
  Arms: Preemptive group

SUMMARY:
Intense e recurrent nociceptive stimulation, which occurs in the postoperatively, can trigger sensitization of the peripheral and central nociceptive pathway, leading to chronic pain. Patients with rotator cuff injury often present to surgery due to referred moderate to intense long-term pain. During the immediate postoperative period, pain is rare due to the routine administration of a brachial plexus blockade as an adjuvant to improve the quality of postoperative analgesia. However, after the second postoperative day, the effect of the blockade ceases, and the pain becomes high and hard to treat, leading the patient to request administration of more frequent and more potent analgesics. The aim of this project is to assess the postoperative analgesic benefits of a brachial plexus blockcade 2 days before arthroscopic surgical correction of rotator cuff injury by reducing the sensitization of the nociceptive pathway.

DETAILED DESCRIPTION:
This is a prospective, controlled, blinded, randomized trial design, based on the PICO structured question: "Brachial plexus block 48 h before arthroscopic surgery for correction of rotator cuff tear in a patient with chronic shoulder pain can influence the postoperative pain? The project will be submitted to the Research Ethics Committee and, after its approval, will be submitted to the Ethics Committee of the institution where the research will be carried out. After approval at these instances and registration at clinicaltrials.gov, a sample of 70 individuals will be selected from a population of patients scheduled for arthroscopic correction of rotator cuff tears. Study subjects will be randomly distributed by electronic draw into two groups: the standard group (SG) and the preemptive group (PG). All patients in both groups will be instructed on the visual analogue (AVS) and numeric pain scales (NPS). The groups will be drawn by a member of the team who will only have the function of controlling the flow of the groups, without participating in any evaluation regarding the trial protocol. All patients in the study will be submitted to BPB and sedation immediately before the surgery. GP patients will undergo BPB 48 h before surgery to try to desensitize the nociceptive pathway. Individuals in the stardard group (SG) will be submitted to an ultrasonographic examination of the topography of the shoulder to be operated on, without knowing whether any therapeutic procedure was performed or just an examination. Both components of both groups will be instructed to use a sling after the procedure 48 h before surgery (BPB or US exam).

INCLUSION CRITERIA: patients scheduled for arthroscopic correction of rotator cuff injury, body mass index < 35 kg/m², shoulder pain complaint for at least 3 months and intensity ≥ 4 (0 to 10) on the day of the pre-anesthetic consultation , ASA I or II, mental and legal capacity to spontaneously accept and sign the informed consent form.

EXCLUSION CRITERIA: allergy to any drug in the study protocol, refusal to participate, contraindication to any substance or technique described in the protocol, intellectual or other limitations that make it difficult to understand the questions and guidelines related to the project protocol, intercurrence at the time of the BPB, not properly installing the BPB (assessment of its sensory effect).

SAMPLE SIZE. The authors carried out an unpublished study comparing two groups of 30 patients for arthroscopic correction of cuff injuries under BPB guided by a peripheral nerve stimulator associated with general anesthesia. One group received BPB 2 days before surgery to assess the possible advantage of reducing the sensitization of chronically stimulated nociceptive pathways in reducing postoperative pain. It is known that postoperative pain in this scenario becomes more intense from the third day on. In this study, pain on the third postoperative night had a mean score of 3.68 (END - 0 to 10), with a standard deviation of 3.04. Our goal is to reduce scores below 3 on the third postoperative night (we will consider an average of 2). Using Pocock's formula12, for a significance level of 95% and a statistical power of 80%, the calculated sample size was 25.86. We increased it to 35 to compensate for losses, with a total of 70 patients in the study.

TECHNIQUE. After guidance on the protocol and signature of the TCLE (Annex 1), the 70 individuals from the study sample will be randomly distributed into two groups (preemptive group - PG; standard group - SG) using an electronic draw offered on the website www.random.org. After distributing the numbers, the same professional responsible for it will number 70 brown envelopes from 1 to 70 and inside each one of them will put the name of the group that corresponds to it, according to the order established by the draw. The order of arrival of patients at the pre-anesthetic evaluation office will correspond to the order in which the envelopes are numbered. The professional responsible for drawing lots and distributing envelopes will not participate in anesthesia or evaluations and will keep the draw secret for security and any clarifications. In the pre-anesthetic consultation, patients with shoulder pain for more than 3 months and with a pain score on the day of the consultation ≥ 4 who agreed to participate in the study will respond to the brief pain inventory validated for Brazilian Portuguese13, to the short version of the questionnaire McGill's pain test14 and the quality of life questionnaire validated for Brazilian Portuguese (WHOQOL-SRPB)15.

After basic monitoring (electrocardioscopy - ECG, oximetry and non-invasive blood pressure - NIBP) and obtaining venous access, PG patients will receive BPB 48 h before surgery. The BPBs in the study will be US-guided. In preemptive BPB (PG), 15 ml of 1% ropivacaine will be injected. Patients in the SG will be submitted to an ultrasound examination of the brachial plexus, and even if they are not submitted to a puncture or invasive process, they will not know which group they will participate in to keep them covered. The anesthesiologist who performs the previous BPB may be the same one who will perform the BPB for that patient on the day of the surgery, since the mark of the first BPB will hardly have disappeared, making it practically impossible to cover up this sign. Likewise, the anesthesiologist who will perform the previous ultrasound examination may be the same one who will perform the BPB on the day of the surgery. All patients in both groups will be instructed to use a sling on the shoulder to be operated after the previous BPB or previous ultrasound examination, in an attempt to keep the group covered. The anesthesiologist conducting the sedation and assessment of patients will not be able to participate in the blocks or examination of the patient who will be administering the sedation or performing the assessment. Patients will be instructed to use dipyrone 1 g every 6 hours and paracetamol (500 mg) associated with codeine (30 mg) in case of pain ≥ 4 in the two days prior to surgery. On the day of surgery, all patients will be asked about the intensity of pain at that time (record). After that, patients in both groups will undergo basic monitoring (as mentioned above) upon entering the operating room, obtaining venous access, sedation with 3 mg of midazolam and fentanyl 50 µg, and BPB with the same technique and block material preemptive. After confirming the installation of the BPB, the patient will receive intravenous ketamine 15 mg. The adjuvant medication will be dipyrone 30 mg/kg, cephalozine 2 g, ketoprofen 100 mg, ondansetron 8 mg, dexamethasone 4 mg. Hemodynamic changes will be managed at the discretion of the providing anesthetist.

It is routine for the team to perform surgeries in the morning and to discharge patients in the late afternoon, except for exceptions due to intercurrences. In the postoperative period, all patients will receive dipyrone 1 g every 6 hours and the combination of paracetamol (500 mg) and codeine (30 mg) as rescue for postoperative pain ≥ 4.

All patients will receive telephone contact from the evaluator between 5:00 pm and 7:00 pm of the first three postoperative days, when they will respond when the first pain ≥ 4 occurred in the postoperative period, what is the consumption of paracetamol/codeine. In the first two days, the level of pain at the time of the interview and the average pain during the day will be recorded. On the third day, patients will answer the brief pain inventory questionnaire13, the McGill pain questionnaire14 and the quality of life questionnaire (WHOQOL)15

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 35 kg/m²
* shoulder pain lasting > 3 months
* pain score > 3 (visual analog scale and verbal response 0 to 10) on the day of pre anesthetic evaluation
* American Society of Anesthesiologists score I or II
* mentally and legally capable to understand and consent to study participation.

Exclusion Criteria:

* Allergy to any medication of the trial
* refusal to participate, contraindication to any medication or technique described in the protocol of the trial
* complications from, or failure of brachial plexus blockade.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Pain score on third postoperative day | Three days
  Pain assessment through verbal numerical scale of pain (from 0 to 10).

SECONDARY OUTCOMES:
Pain scores before surgery. | Just before surgery
  Postoperative pain through verbal numerical scale of pain (from 0 to 10)
Pain cores on three postoperative days. | Three days.
  Postoperative pain through verbal numerical scale os pain (from 0 to 10)
Opioid consumption | Two days before surgery
  Opioid consumption (mg codeine) two days before surgery
Opioid consumption | Three days
  Opioid consumption (mg codeine) during the first three postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Vieira, Professor, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will only be available for researchers after the end of the data collection and analysis on request.